CLINICAL TRIAL: NCT01243892
Title: A Phase IV, Open Label, Multicenter, Case-controlled Study of Growth in Patients Using the Nutropin AQ® Nuspin®
Brief Title: A Study to Evaluate Growth in Participants Treated With Somatropin (Nutropin) Using NuSpin Device
Status: Terminated | Type: Observational
Why Stopped: The study was closed due to the slow enrollment rate.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: L4917g; ML01311 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone; Growth Hormone; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1: IGHD participants: Isolated growth hormone deficient (IGHD) participants who initiated somatropin (Deoxyribonucleic acid [DNA] origin) (recombinant human growth hormone [rhGH]) using the NuSpin device, will be observed for at least 2 years. The choice of initiation of NuSpin treatment and the treatment regimen will be as per treating physician's discretion, the study protocol does not enforce or specify any treatment regimen.
  Interventions: Device: NuSpin; Drug: Somatropin
- Cohort 2: ISS participants: Idiopathic short stature (ISS) participants who initiated somatropin (DNA origin) (rhGH) using the NuSpin device, will be observed for at least 2 years. The choice of initiation of NuSpin treatment and the treatment regimen will be as per treating physician's discretion, the study protocol does not enforce or specify any treatment regimen.
  Interventions: Device: NuSpin; Drug: Somatropin

INTERVENTIONS:
Device: NuSpin — Device for administration of doses of somatropin.
Drug: Somatropin — Somatropin using either NuSpin or Nutropin AQ Pen, as per standard dosing.
  Other Names: Nutropin AQ (Somatropin [DNA Origin] injection)

SUMMARY:
This is a Phase IV, open label, case-controlled, observational study to evaluate the age-adjusted cumulative height velocity in pre-pubertal isolated growth hormone deficient (IGHD) and idiopathic short stature (ISS) participants receiving daily doses of somatropin (recombinant human growth hormone [rhGH]; Nutropin) using NuSpin device compared to historical controls from the national cooperative growth study (NCGS).

ELIGIBILITY:
Inclusion Criteria:

* Bone age less than or equal to (</=) 8 years (females) or </= 10 years (males) as determined by x-ray of the left hand and wrist obtained within six months before enrollment
* Prepubertal males and females by physical exam
* Naive to rhGH therapy
* Diagnosis of IGHD or ISS by standard pharmacologic testing and no other discernable etiology for short stature
* Height standard deviation score (Ht SDS) </= -1.5 (</= 5th percentile) for IGHD participants; Ht SDS </= -2.25 (</= 1.2 percentile) for ISS participants

Exclusion Criteria:

* Short stature etiologies other than IGHD or ISS
* Participants receiving chronic corticosteroid therapy (greater than [>] 3 months) for other medical conditions
* Participants with active malignancy or any other condition that the investigator believes would pose a significant hazard to the participant if rhGH were initiated
* Females with turner syndrome
* Any previous rhGH treatment
* Participation in another simultaneous medical investigation or trial
* Pediatric participants with closed epiphyses
* Participants prescribed rhGH doses outside the variance of NCGS control participant dosing

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Somatropin-naive pre-pubertal participants with growth hormone deficiency or ISS
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Aaron Davis, M.D., Study Director — Genentech, Inc.
Locations (14):
- United States (14):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Sacramento, California
  - San Diego, California
  - Greenwood Village, Colorado
  - Palm Bay, Florida
  - Pembrook Pines, Florida
  - Atlanta, Georgia
  - Wheaton, Illinois
  - Minneapolis, Minnesota
  - Mount Kisco, New York
  - New Rochelle, New York
  - Columbus, Ohio
  - Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to slow enrollment, the study was terminated after screening 33 participants and enrolling only 18 participants, out of 480 planned participants.
Groups:
- IGHD Participants: Isolated growth hormone deficient (IGHD) participants who initiated somatropin (Deoxyribonucleic acid [DNA] origin) (recombinant human growth hormone [rhGH]) using the NuSpin device, were observed for at least 2 years. The choice of initiation of NuSpin treatment and the treatment regimen was as per treating physician's discretion, the study protocol did not enforce or specified any treatment regimen.
- ISS Participants: Idiopathic short stature (ISS) participants who initiated somatropin (DNA origin) (rhGH) using the NuSpin device, were observed for at least 2 years. The choice of initiation of NuSpin treatment and the treatment regimen was as per treating physician's discretion, the study protocol did not enforce or specified any treatment regimen.
Period: Overall Study
Arm/Group | IGHD Participants | ISS Participants
Started | 15 | 3
Completed | 13 | 3
Not Completed | 2 | 0
Not completed — Did not meet eligibility criteria | 2 | 0

BASELINE CHARACTERISTICS:
Population: Study population included all enrolled somatropin-naive pre-pubertal participants with growth hormone deficiency or ISS.
Groups:
- IGHD Participants: IGHD participants who initiated somatropin (DNA origin) (rhGH) using the NuSpin device, were observed for at least 2 years. The choice of initiation of NuSpin treatment and the treatment regimen was as per treating physician's discretion, the study protocol did not enforce or specified any treatment regimen.
- ISS Participants: ISS participants who initiated somatropin (DNA origin) (rhGH) using the NuSpin device, were observed for at least 2 years. The choice of initiation of NuSpin treatment and the treatment regimen was as per treating physician's discretion, the study protocol did not enforce or specified any treatment regimen.
- Total: Total of all reporting groups
Arm/Group | IGHD Participants | ISS Participants | Total
Number analyzed (Participants) | 15 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.60 (2.07) | 8.11 (2.60) | 9.35 (2.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 13 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Annualized Height Velocity in Response to rhGH Treatment Using the NuSpin Device After Two Years of Treatment
Description: The annualized height velocity (cm per year [cm/yr]) over 2 years was calculated as: [(height in cm at t24 minus (-) height in cm at t0) divided by (date at t24 - date at t0)] multiplied by 365.25, where, t0 is the baseline measurement visit and t24 is the 2-year measurement visit.
Time Frame: Baseline up to Month 24 (Year 2)
Population: Data for this outcome measure was not collected as the study was terminated prematurely due to slow enrollment.
Arm/Group | IGHD Participants | ISS Participants
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Annualized Height Velocity in Response to rhGH Treatment Using the NuSpin Device for First Year of Treatment
Description: The annualized height velocity (cm/yr) after 1 year was calculated as: [(height in cm at t12 - height in cm at t0) divided by (date at t12 - date at t0)] multiplied by 365.25, where, t0 is the baseline measurement visit and t12 is the 1-year measurement visit.
Time Frame: Baseline up to Month 12 (Year 1)
Population: Data for this outcome measure was not collected as the study was terminated prematurely due to slow enrollment.
Arm/Group | IGHD Participants | ISS Participants
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Annualized Height Velocity in Response to rhGH Treatment Using the NuSpin Device During the Second Year of Therapy
Description: The annualized height velocity (cm/yr) for second year was calculated as: [(height in cm at t24 - height in cm at t12) divided by (date at t24 - date at t12)] multiplied by 365.25, where, t12 is the 1-year measurement visit and t24 is the 2-year measurement visit.
Time Frame: Month 12 to Month 24 (Year 1 to Year 2)
Population: Data for this outcome measure was not collected as the study was terminated prematurely due to slow enrollment.
Arm/Group | IGHD Participants | ISS Participants
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 9 months
Description: Study population included all enrolled somatropin-naive pre-pubertal participants with growth hormone deficiency or ISS.
Arm/Group | IGHD Participants | ISS Participants
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/3
Other Adverse Events (participants affected / at risk) | 0/15 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGHD Participants (N=15) | ISS Participants (N=3)
Peripheral oedema (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGHD Participants (N=15) | ISS Participants (N=3)
Gastroenteritis (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.